CLINICAL TRIAL: NCT03930602
Title: An Open-label, Single-sequence Study to Investigate the Effects of Cytochrome P450 1A2 Inhibition on the Pharmacokinetics of BMS-986165 in Healthy Participants
Brief Title: Study to Characterize the Effects of Cytochrome p450 1A2 Inhibition on Systemic Exposure to BMS-986165
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IM011-088
Record Dates: First submitted 2019-04-26; First posted 2019-04-29 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — deucravacitinib; Fluvoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986165+Fluvoxamine (Experimental)
  Interventions: Drug: BMS-986165; Drug: Fluvoxamine
- BMS-986165 only (Experimental)
  Interventions: Drug: BMS-986165
- Fluvoxamine only (Experimental)
  Interventions: Drug: Fluvoxamine

INTERVENTIONS:
Drug: BMS-986165 — Participants will receive BMS-986165.
  Arms: BMS-986165 only; BMS-986165+Fluvoxamine
Drug: Fluvoxamine — Participants will receive fluvoxamine.
  Arms: BMS-986165+Fluvoxamine; Fluvoxamine only

SUMMARY:
To compare the pharmacokinetic characteristics of BMS-986165 after a single-dose administration alone vs. in combination with fluvoxamine (CYP1A2 inhibitor)

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant, as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations in the opinion of the investigator.
* Body mass index of 18 to 32 kilograms per square meter (kg/m2), inclusive, and body weight ≥ 50 kg, at screening.
* Normal renal function at screening as evidenced by an estimated glomerular filtration rate (GFR) > 80 milliliter/minute/1.732 meter square calculated with the Chronic Kidney Disease Epidemiology Collaboration formula.

Exclusion Criteria:

* Any significant acute or chronic medical condition that presents a potential risk to the participant and/or may compromise the objectives of the study,
* Any major surgery within 4 weeks of study drug administration
* Participants who currently smoke, as well as those who have stopped smoking less than 6 months prior to dosing on Day 1.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986165 | 10 days
AUC(0-T) of BMS-986165 | 10 days
AUC(INF) of BMS-986165 | 10 days

SECONDARY OUTCOMES:
Fluvoxamine steady-state plasma concentrations | 10 days
Percentage of participants with Adverse events (AEs) | From screening up to end of drug treatment (Day 13)
Percentage of participants with Serious Adverse events (SAEs) and Death | From screening up to end of drug treatment (Day 13)
Percentage of participants with Adverse events (AEs) leading to discontinutation | From screening up to end of drug treatment (Day 13)
Percentage of participants with clinical significant laboratory abnormalities vital sign measurements and ECGs | From screening up to end of drug treatment (Day 13)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- ICON Plc (PRA Health Sciences), Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm